CLINICAL TRIAL: NCT04359628
Title: How Does Patients' Overall Assessment of Their Health Vary Across and Within Different Disease Groups? A Study Protocol to Study Health-related Quality of Life Using the EQ-5D in the Swedish National Quality Registers
Brief Title: How Does Patients' Overall Assessment of Their Health Vary Across and Within Different Disease Groups?
Acronym: SWEQR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Karolinska Institutet (Other); Linkoeping University (Other Government); Lund University (Other); Ryhov County Hospital (Other); Göteborg University (Other); Umeå University (Other); University of Melbourne (Other); Office of Health Economics, London (Unknown)
Responsible Party: Principal Investigator, Ola Rolfson, Professor, Vastra Gotaland Region
Other Study IDs: 1185-18/2019-00812
Record Dates: First submitted 2020-04-15; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Hip Disease; Heart Failure; Psoriasis; Fractures, Bone; Bipolar Disorder; Respiratory Failure; Knee Disease; Knee Injuries; Ankle Disease; Spinal Disease; Rheumatic Diseases; Osteoarthritis
Keywords: health-related quality of life; quality register; EQ-5D; patient-reported outcomes; patient-reported outcome measures; comorbidity; EQ VAS; experience-based values; health state valuation; hypothetical values; patient values
MeSH Terms: conditions — Heart Failure; Psoriasis; Fractures, Bone; Bipolar Disorder; Respiratory Insufficiency; Knee Injuries; Spinal Diseases; Rheumatic Diseases; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (13):
- BOA: Patients with osteoarthritis registered in the Better BOA register
- Swedankle: Patients who underwent ankle replacement, fusion or osteotomies and registered in the Swedish ankle registry
- xBase: Patients with cruciate ligament injuries who received surgical treatment and were registered in the Anterior Cruciate Ligament Register
- SFR: Patients who received treatment in the Swedish Fracture Register
- SHAR: Patients who underwent hip replacement therapy and registered in the Swedish Hip Arthroplasty Register
- SKAR: Patients with knee osteoarthritis and other diagnoses who underwent knee replacement or osteotomies and were registered in the Swedish Knee Arthroplasty Register
- Bipolär: Patients with Bipolar disorder receiving treatment and were registered in the Swedish National Register for Bipolar Disorder
- Swedevox: Patients with respiratory failure receiving technical respiratory assistance and were registered in the Swedish National Registry for Respiratory Failure
- PsoReg: Patients receiving systemic treatment for psoriasis and were registered in the Swedish Registry for Systematic Psoriasis Treatment
- SRQ: Patients with rheumatic disease receiving medical treatment and rehabilitation and were registered in the Swedish Rheumatology Quality Register
- SwedeHF: Patients who received treatments of different types in the Swedish Heart Failure Registry
- Swespine: Patients with spinal stenosis, disc hernia and related diagnoses receiving surgical spine treatment and were registered in the Swedish Spine Register
- Population health survey: Data of members of the general population who answered population surveys using the EQ-5D-3L instrument

SUMMARY:
EQ-5D is one of the most commonly employed patient-reported outcome (PRO) measures. It is included in many of the Swedish National Quality Registers (NQRs). EQ-5D health states are usually summarized using 'values' obtained from healthy members of the general public. However an alternative - which remains to be studied in detail - is the potential to use patients' self-reported overall health on the visual analogue scale as a means of capturing experience-based values. The overall aim of this project is to increase knowledge on the potential applicability of EQ VAS as a health state valuation method through assessment of its variability across and within patient groups and compared with that of the general population in Sweden.

Data on nearly 700,000 patients from 12 NQRs covering a variety of diseases/conditions and from the general population will be analysed. Longitudinal studies of PROs among different patient groups will be conducted at baseline/first visit and 1-year follow-up. Descriptive analyses comparing EQ-5D health states and observed self-assessed EQ VAS within and across registers will be performed. Comparisons of the change in health state and observed EQ VAS values over one year will also be made. Regression models will be used to assess whether EQ-5D dimensions predict observed EQ VAS values to investigate patient value sets in each NQR. These will be compared across the patient groups and with the existing Swedish experience-based VAS and time trade-off (TTO) value sets obtained from the general population. This research project will provide information on the variation among different patient groups in terms of self-reported health status through EQ VAS and comparison with the general population. Knowledge on the relative importance of different dimensions of the EQ-5D to different patient groups as well as the general population will be gained in this project. The possibility of getting value sets based on patients' self-reported EQ VAS values and their comparison with value sets from experience-based general population studies will be discussed.

DETAILED DESCRIPTION:
Research questions:

1. How do EQ-5D health states and self-assessed EQ VAS values vary across and within patient groups, and over follow-up stages, and in comparison to the general population data?
2. To what extent do EQ-5D health states predict EQ VAS values, and how do the resulting experience-based patient value sets differ when estimated from patients' data at baseline and 1-year follow-up and how do the EQ VAS values predicted for EQ-5D health states differ between different patient groups?
3. How do these patient value sets modelled using data from the registers compare with the Swedish VAS and TTO experience-based EQ-5D value sets obtained from the general population?
4. How do value sets for EQ-5D-3L, predicted from EQ VAS differ from value sets predicted for the EQ-5D-5L, predicted from its EQ VAS?

Data: In this project 12 National Quality Registries holding records of PROs, on the EQ-5D instrument, records of approximately 700,000 patients will be included. Clinical data (age, sex, BMI, diagnosis (es) and interventions) and PROs data (EQ-5D-3L and condition-specific) will be retrieved from the registries. Data from cross-sectional population surveys in Sweden will be included for comparison; a total of approximately 45,000 records used in developing the Swedish TTO and VAS value sets.

The quality registries to be part of the study include;

1. Better management of patients with osteoarthritis (BOA)
2. The Swedish Ankle Registry (Swedankle)
3. The Swedish Fracture Register (SFR)
4. The Swedish Heart Failure Registry (SwedHF)
5. The Swedish Hip Arthroplasty Register (SHAR)
6. The Swedish Knee Arthroplasty Register (SKAR)
7. The Swedish National Anterior Cruciate Ligament Register (XBase)
8. The Swedish National Quality Register for Bipolar Disorder (BipoläR)
9. The Swedish National Registry for Respiratory Failure (Swedevox)
10. The Swedish Registry for Systematic Psoriasis Treatment (PsoReg)
11. The Swedish Rheumatology Quality Register (SRQ)
12. The Swedish Spine Register (Swespine)

Data analysis: Records of patients in the registries with baseline and follow-up data on PROs will be included for the different analyses to be conducted. The analyses will focus on the three main data components coming from the EQ-5D instrument. Data collected by the EQ-5D descriptive system on the five dimensions; the EQ-VAS score and EQ-5D index resulting from transforming the EQ-5D health profile into a single index using value sets. Hence, analyses looking into how the EQ-5D profile varies within and across patient groups and how it varies over time will form one component of the analyses to be conducted. Similarly, the pattern of EQ-VAS scores across patient groups and follow-ups will be analysed. Similar comparisons of EQ-5D index within and across patient groups, based on current Swedish value sets and patient VAS value sets to be elicited from the dataset, will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at baseline/first visit registration
* Completed the PRO instrument, EQ-5D, at least at the baseline /first visit

Exclusion Criteria:

* Incomplete data on age, sex, or EQ-5D dimensions

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes patients who received medical, surgical and/or other related treatments and were registered in one of the 12 National Quality Registries (NQRs) in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 700000 (Estimated)
Dates: Start 2002-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Problems reported on the EQ-5D dimensions (EQ-5D-3L and EQ-5D-5L) | At baseline/ first visit
  These describe the proportions of levels of problems reported in each of the EQ-5D-3L or EQ-5D-5L dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression)
Problems reported on the EQ-5D dimensions (EQ-5D-3L and EQ-5D-5L) | At 1-year follow-up
  These describe the proportions of levels of problems reported in each of the EQ-5D-3L or EQ-5D-5L dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression)
EQ-VAS value | At baseline/ first visit
  It describes an overall assessment by respondent of their health, ranging on a scale from 0 (worst imaginable health) to 100 (best imaginable health).
EQ-VAS value | At 1-year follow-up
  It describes an overall assessment by respondent of their health, ranging on a scale from 0 (worst imaginable health) to 100 (best imaginable health).
EQ-5D index (for EQ-5D-3L and EQ-5D-5L) | At baseline/ first visit
  An index calculated from the five EQ-5D (3L and 5L) dimensions by attaching specific weights to each severity level in each dimension.
EQ-5D index (for EQ-5D-3L and EQ-5D-5L) | At 1-year follow-up
  An index calculated from the five EQ-5D (3L and 5L) dimensions by attaching specific weights to each severity level in each dimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Registercentrum, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teni FS, Rolfson O, Devlin N, Parkin D, Naucler E, Burstrom K; Swedish Quality Register (SWEQR) Study Group. Longitudinal study of patients' health-related quality of life using EQ-5D-3L in 11 Swedish National Quality Registers. BMJ Open. 2022 Jan 6;12(1):e048176. doi: 10.1136/bmjopen-2020-048176. PMID 34992101
- [Derived] Teni FS, Rolfson O, Devlin N, Parkin D, Naucler E, Burstrom K; Swedish Quality Register (SWEQR) Study Group. Variations in Patients' Overall Assessment of Their Health Across and Within Disease Groups Using the EQ-5D Questionnaire: Protocol for a Longitudinal Study in the Swedish National Quality Registers. JMIR Res Protoc. 2021 Aug 27;10(8):e27669. doi: 10.2196/27669. PMID 34448726